CLINICAL TRIAL: NCT04984239
Title: Adapting Acceptance and Mindfulness-based Behavior Therapy for Stroke Survivors With Aphasia to Improve Communication Success, Post-stroke Adaptation, and Quality of Life
Brief Title: Adapting Acceptance and Commitment Therapy for Stroke Survivors With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Delaware (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, William Evans, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20090213; R03HD104246-01 (NIH)
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Aphasia
Keywords: Counseling; Therapeutics
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy adapted for aphasia (Other): There is only a single study arm, in which the adapted intervention will be developed using a successive cohort design.
  Interventions: Behavioral: Acceptance and Commitment Therapy for aphasia

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for aphasia — The intervention will consist of Acceptance and Commitment Therapy modified to meet the needs of stroke survivors with aphasia, combined with communication strategy training.

SUMMARY:
The proposed study is a Stage I successive cohort trial intended to adapt Acceptance and Commitment Therapy (ACT) to meet the specific needs of stroke survivors with aphasia ("ACT for Aphasia"). It will do so by incorporating communication supports and compensatory speech-language treatment. The goal of developing this integrated treatment is to improve successful communication participation, psychosocial adjustment, and quality of life for stroke survivors with aphasia.

In the first phase of the project, the investigators will create a treatment manual with input from a stakeholder advisory board consisting of caregivers and stroke survivors with aphasia. The investigators will then recruit an initial cohort of five stroke survivors with aphasia to undergo the initial version of the treatment based and provide feedback. This will aid revision of the manual, which the investigators will then evaluate using a second cohort of 16 stroke survivors with aphasia. The investigators predict that ACT for Aphasia will be acceptable and feasible based on measures of participant satisfaction and treatment adherence. The investigators will also measure pre- to post-treatment changes in psychological distress, functional disability, quality of life, and communication participation and functioning to establish preliminary effect size estimates for this intervention, in preparation for a subsequent Stage II efficacy trial.

DETAILED DESCRIPTION:
The overarching goals of this research are to improve psychosocial adjustment, quality of life, and successful communication participation by developing Act for Aphasia, a patient-centered, manualized behavioral intervention in Stage I research. Stroke survivors with aphasia will complete a 10-session intervention. In study Aim 1, the investigators will engage a Stakeholder Advisory Board (SAB) of people with aphasia (PWA) and caregivers to provide input to develop a treatment manual. The investigators will then use an iterative design process and two successive participant cohorts to refine the manual. Cohort 1 (N=5) will participate in the initial version of the treatment, then help inform its revision by being invited to join the SAB. Cohort 2 (N=16) will participate in the revised version. In Aim 2a the investigators will establish feasibility and acceptability of this intervention. In Aim 2b the investigators will estimate preliminary effect sizes for a subsequent Stage II efficacy trial.

Participant assignment: given the early phase of this research and the lack of control conditions or groups, there will be no random assignment. Participants will be enrolled in the study as they are referred and found to be eligible, with the first five participants being enrolled in the first study cohort during year 1 while the remainder of participants will be enrolled in the second cohort across years 1 and 2.

Intervention description: the ACT for Aphasia treatment manual will be a 10-session intervention created by modifying an existing ACT manual provided by Dr. Meyer. To meet the specific needs of stroke survivors with aphasia, ACT will be modified in two main ways. First, the intervention will include modified language and communication supports to address the unique communication challenges faced by people with aphasia that could impede engagement with ACT content. Multi-modality communication supports will be provided by the treating clinician (e.g., writing out key words to support verbal content, summarizing and providing repetitions, providing session summaries to review between sessions). Manual creation will follow existing practice recommendations for modifying counseling interventions for PWA (e.g., simplifying language and increasing use of visual metaphors) which will be reviewed by the SAB. Second, ACT will be further augmented via individualized language compensation training and a focus on identifying and addressing communication-based barriers to life participation. Language training will focus on active compensatory strategies such as self-cuing, use of alternative modalities (gesture, writing), and use of commonly available technology (e.g., smartphone dictionaries, text-to-speech). The details of this language compensation training will also be determined based on input from the SAB, and will be revised after reviewing performance and interview feedback from each successive cohort.

Intervention administration procedures: all aspects of the treatment protocol will be administered by Dr. Evans or a licensed speech-language pathologist on study staff who has received training in providing ACT. The intervention will consist of 10 weekly treatment sessions. Post-treatment interviews providing feedback for protocol revision will be administered by Dr. Evans within 2 weeks of study completion. Interviews will use a semi-structured, ethnographic interview approach and be video-recorded. These interviews will ask specific questions about the participant's experience and perspective regarding each functional domain of the intervention (i.e., the "Open Up," "Be Present," and "Do What Matters" components of ACT and the individualized language compensation training), and will be asked for suggestions and improvements about the specific content and techniques employed.

Note that the values tracker measure was formally removed from the outcome measures in the study protocol. The protocol was modified to administer the values tracker informally during the treatment phase to help clinicians monitor progress and to guide in-session treatment discussions about value-based goal setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be age 18 or older.
* Participants will have an existing diagnosis of aphasia subsequent to left hemisphere stroke.

Exclusion Criteria:

* Participants with a history of other acquired or progressive neurological disease.
* Participants whose mean modality t-score falls below 40 on the spoken language comprehension subdomain of the Comprehensive Aphasia Test.
* Participants with semantic memory impairments as determined by the cutoff of the semantic memory component of the Comprehensive Aphasia Test.
* Participants with unmanaged drug /alcohol dependence.
* Participants with severe diagnose.d mood or behavioral disorders that require specialized mental health interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Evans, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Language Rehab and Cognition Lab, Department of Communication Sciences and Disorders, School of Health and Rehabilitation Sciences, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this research will be shared with the wider scientific community in a timely fashion, concurrent with publication with no planned end date. Materials shared in this fashion will consist of all de-identified participant assessment and outcome data, acceptability and feasibility measures, the study protocol, statistical analysis plan, and treatment manual. These materials will be shared via the National Institute of Child Health and Human Development Data and Specimen Hub (NICHD DASH) and made additionally available by sharing the developed treatment manual and other supporting information on Dr. Evans' lab website.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared at the time of study publication without planned end to access.
Access Criteria: Anyone who wishes to access the data.
URL: https://dash.nichd.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study utilized a Stakeholder Advisory Board (SAB) of people with aphasia and care partners to provide input on treatment development. Members of the SAB were not study participants, and therefore were not enrolled as participants.
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Started | 20
Cohort 1 | 5
Cohort 2 | 15
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Scores on the Client Satisfaction Questionnaire - 8
Description: The Client Satisfaction Questionnaire - 8 (CSQ-8) is a brief questionnaire demonstrated to provide "efficient, sensitive, and reasonably comprehensive" measures of patient satisfaction. It has 8 questions rated on a 4-point scale (summed scores range from 8 to 32). High scores indicate high satisfaction and low scores indicate low satisfaction. The CSQ-8 is the primary measure which will determine acceptability of the proposed pilot intervention.
Time Frame: Post-treatment (within one week of completing the treatment phase)
Population: Data from 17 of the 19 completed participants were included in this analysis. This is due to missing data from the remaining 2 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 17
score on a scale | 29.7 (5.3)

2. Secondary Outcome: Mean Scores on the Acceptance and Action Questionnaire II
Description: The Acceptance and Action Questionnaire II (ACQ-II) is a self-report measure of psychological flexibility, acceptance, and experiential avoidance. It has 7 items rated on a 7-point scale (summed scores range from 7 to 49). Higher total scores reflect less psychological flexibility, while lower total scores reflect more flexibility. The ACQ-II will evaluate changes in psychological flexibility, the hypothesized mechanism of action underlying ACT for aphasia.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
score on a scale
  Pre-Treatment | 20.6315789 (9.52313281)
  Post-Treatment | 15.4210526 (8.94002106)

3. Secondary Outcome: Mean Scores on the Acceptance and Action Questionnaire - Acquired Brain Injury
Description: The Acceptance and Action Questionnaire - Acquired Brain Injury (ACQ-ABI) is a 15 item self-report measure adapted from the ACQ-II specifically for people with acquired brain injury based on a 5-point Likert scale ranging from 15-75 where higher scores indicate greater levels of acceptance. While the ACQ-II addresses psychological flexibility generally, the ACQ-ABI measures psychological flexibility relating specifically to the consequences of acquired brain injury and is therefore an informative addition. Similar to the ACQ-II, it will also evaluate changes in psychological flexibility, the hypothesized mechanism of action underlying ACT for aphasia.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
score on a scale
  Pre-Treatment | 49 (8.0346472)
  Post-Treatment | 45.9473684 (9.52466788)

4. Secondary Outcome: Mean Scores on the Kessler K6 Non-specific Distress Scale
Description: The Kessler K6 is a brief, validated instrument that assesses non-specific psychological distress experienced over the past 30 days. It has 6 items rated on a 0 to 4-point scale (summed scores range from 0 to 24). Higher total scores reflect greater psychological distress.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
score on a scale
  Pre-Treatment | 7.26315789 (4.025503492)
  Post-Treatment | 3.84210526 (3.775110858)

5. Secondary Outcome: Mean Scores on the Stroke and Aphasia Quality of Life Scale
Description: The Stroke and Aphasia Quality of Life Scale is a 39-item patient reported measure of qualify of life adapted specifically for people with aphasia from the stroke survivor quality of life scale.
  Total Mean Score: 39 items scored on 1-5 scale Physical Sub-Domain Mean Score: 16 items scored on 1-5 scale Communication Sub-Domain Mean Score: 7 items scored on a 1-5 scale Psychosocial Sub-Domain Mean Score: 16 items scored on 1-5 scale
  For the total score and each subdomain score, values are determined by adding the sum of items relevant to that score (all 39 items for the total mean score, 16 items for the Physical Sub-Domain Mean Score, 7 items for the Communication Sub-Domain Mean Score, 16 items for the Psychosocial Sub-Domain Mean Score), then dividing by the number of relevant items for that score. In each case, the resulting maximum score of 5 and a minimum score of 1, with higher scores indicating higher quality of life.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
score on a scale
  Pre-Treatment Total Mean Score | 3.747789 (0.56973)
  Post-Treatment Total Mean Score | 4.039421 (0.617423)
  Pre-Treatment Physical sub-domain Mean Score | 4.135211 (0.696638)
  Post-Treatment Physical sub-domain Mean Score | 4.148211 (0.88102)
  Pre-Treatment Communication sub-domain Mean Score | 3.270842 (0.800904)
  Post-Treatment Communication sub-domain Mean Score | 3.744368 (0.777438)
  Pre-Treatment Psychosocial sub-domain Mean Score | 3.562737 (0.852164)
  Post-Treatment Psychosocial sub-domain Mean Score | 4.059368 (0.683571)

6. Secondary Outcome: Mean Scores on the Aphasia Outcome Measure
Description: The Aphasia Communication Outcome Measure (ACOM) is a measure of patient-reported "communication functioning," defined as the ability to effectively convey and receive personally relevant messages in natural environments. Results are provided in T scores (sample mean of 50 with a standard deviations of 10), with higher scores indicating better communication functioning.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
T-score
  Pre-Treatment | 55.355625 (8.20934506)
  Post-Treatment | 55.766875 (9.94600806)

7. Secondary Outcome: Mean Scores on the Communication Participation Item Bank
Description: The Communication Participation Item Bank (CPIB) is a patient-reported measure of "communication participation" defined as "taking part in life situations where knowledge, information, ideas or feelings are exchanged." It has been validated for use with community-dwelling adults with multiple different communication disorders, including aphasia. Results are provided in T scores (sample mean of 50 with a standard deviations of 10), with higher scores indicating better communication participation.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 19
T-score
  Pre-Treatment | 45.3052632 (6.78392493)
  Post-Treatment | 47.4105263 (6.06464204)

8. Secondary Outcome: Mean Scores on Modified University of Washington Resilience Scale
Description: The UWRS is a patient-reported outcome measure intended to measure an individual's perceived resilience. The original UWRS has been modified for people with aphasia (mUWRS), and was added to the study protocol for the second cohort of study participants to measure resilience pre- and post-treatment.
  This measure is reported as a T-score with a mean of 50 and a standard deviation (SD) of 10. A higher T-score represents a higher level of resilience.
Time Frame: Baseline and Post-Treatment (within one week of completing the treatment phase)
Population: This outcome measure was used in the second participant cohort only - data from all 14 participants in the second cohort were analyzed.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
Number analyzed (Participants) | 14
T-score
  Pre-Treatment | 48.87143 (11.35439)
  Post-Treatment | 54.10714 (10.149)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of the study, for a total of 14 months.
Arm/Group | Acceptance and Commitment Therapy Adapted for Aphasia
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT04984239/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04984239/SAP_001.pdf
  • Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT04984239/ICF_002.pdf